CLINICAL TRIAL: NCT01979172
Title: Comparison of Intraocular Lens Power Calculation Methods After Corneal Laser Refractive Surgery in Axial and Refractive Ammertropia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The National Eye Hospital, Cairo, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed El Bahrawy, Dr., The National Eye Hospital, Cairo, Egypt
Other Study IDs: LASIK/IOL
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Cataract; Refractive Errors
Keywords: LASIK; Intraocular lens; Biometry; IOL master
MeSH Terms: conditions — Cataract; Refractive Errors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study aims at determining the best biometry calculation formula to be used in IOL calculation of cataract patients how previously underwent laser refractive correction surgery

DETAILED DESCRIPTION:
Patients undergoing laser refractive surgery will will be investigated in means of Pentacam testing and IOL master biometry both preoperative and 6 weeks postoperative to determine which IOL calculation formula is the nearest and most accurate to preoperative records in different refractive sittings.

ELIGIBILITY:
Inclusion Criteria:

* all patient undergoing laser refractive surgery

Exclusion Criteria:

* previous ophthalmic surgery
* previous trauma
* ocular pathology other than refractive error

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient undergoing laser refractive surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Best Selected IOL calculation formula | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rami R Fikry, MD/FRCS, Principal Investigator — Watany Eye Hospital; Ahmed Assaf, MD/FRCS, Study Director — Watany Eye Hospital; Ahmed Osama, MS, Principal Investigator — Watany Eye Hospital; Moahmed O El Bahrawy, MS, Principal Investigator — Watany Eye Hospital
Locations (1):
- Watany Eye Hopsital, Cairo, Cairo Governorate, Egypt

REFERENCES:
- See also: Watany Eye Hospital Official website — http://www.alwatany.net.eg